CLINICAL TRIAL: NCT02809170
Title: The Effect of Arginine and Citrulline Supplementation on Endothelial Dysfunction in Mitochondrial Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tawam Hospital (Other)
Responsible Party: Principal Investigator, Ayman El-Hattab, Consultant, Genetics and Metabolic, Tawam Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CED 343-14
Record Dates: First submitted 2016-06-15; First posted 2016-06-22 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Arginine; Citrulline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arginine (Active Comparator): Endothelial function will be assessed before and after arginine supplementation
  Interventions: Dietary Supplement: Arginine
- Citrulline (Active Comparator): Endothelial function will be assessed before and after citrulline supplementation
  Interventions: Dietary Supplement: Citrulline

INTERVENTIONS:
Dietary Supplement: Arginine — Arginine is an amino acids
  Arms: Arginine
Dietary Supplement: Citrulline — Citrulline is an amino acid
  Arms: Citrulline

SUMMARY:
Mitochondrial diseases occur due to inadequate energy production. In addition, nitric oxide (NO) deficiency occurs in mitochondrial diseases. The endothelial layer of blood vessels functions in maintaining blood vessels patency through producing NO which relaxes vascular smooth muscles and therefore maintains the patency of blood vessels and adequate blood perfusion. In mitochondrial diseases, endothelial cells fail to perform their normal function in maintaining the patency of blood vessels (endothelial dysfunction) because of the inability to produce enough NO. Endothelial dysfunction results in decreased blood perfusion in different organs which can contribute to the complications seen in mitochondrial diseases. The amino acids arginine and citrulline act as NO precursors and can increase NO production. In this study we hypothesize that due to the inability to produce enough NO patients with mitochondrial diseases have endothelial dysfunction that will improve after arginine or citrulline supplementation. The investigators will assess endothelial function using peripheral arterial tonometry before and after arginine or citrulline supplementation. The investigators expect that arginine and citrulline supplementation will improve endothelium function. This will support the therapeutic use of arginine and citrulline in mitochondrial diseases.

DETAILED DESCRIPTION:
The investigators will study 10 children with mitochondrial diseases and 10 healthy control children. The investigators will study control children to be able compare the results of children with mitochondrial diseases to control healthy children. Therefore, the investigators will study control children only once to compare these results to the results of children with mitochondrial diseases at baseline. To assess the effect of arginine and citrulline on children with mitochondrial diseases, the investigators need to assess children with mitochondrial diseases four times. First time as baseline. Then children with mitochondrial diseases will be randomized to receive either oral arginine or citrulline at a dose of 500 mg/kg/day divided in 3 doses daily for 2 weeks after which a second assessment will be performed. Oral arginine or citrulline will be discontinued and after a two-week washout period another baseline assessment will be done. After that, the child will be started on oral citrulline (if the participant received arginine the first time) or arginine (if the participant received citrulline the first time) at a dose of 500 mg/kg/day divided in 3 doses daily for 2 weeks after which a fourth assessment will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of mitochondrial disease with multi-organ disease involving neurological and/or muscular systems.
2. The diagnosis must be confirmed either molecularly (identifying mutations known to be associated with mitochondrial diseases) or by respiratory chain assay abnormalities.

Exclusion Criteria:

1. Have acute illness or physical disability interfering with ability to undergo the study procedures.
2. Known to have other factors that are known to result in endothelial dysfunction including hypertension, hyperlipidemia, and diabetes.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Reactive hyperemic index (RHI) | 2 year
  Reactive hyperemic index (RHI) which reflects endothelial function will be measured using the EndoPAT instrument

SECONDARY OUTCOMES:
Plasma concentration levels of arginine and citrulline | 2 year
  Plasma arginine and citrulline levels will also be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ayman W El-Hattab, MD, Principal Investigator — Tawam Hospital
Locations (1):
- Tawam Hospital, Al Ain City, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes